CLINICAL TRIAL: NCT02332668
Title: A Phase I/II Study of Pembrolizumab (MK-3475) in Children With Advanced Melanoma or a PD-L1 Positive Advanced, Relapsed or Refractory Solid Tumor or Lymphoma (KEYNOTE-051)
Brief Title: A Study of Pembrolizumab (MK-3475) in Pediatric Participants With an Advanced Solid Tumor or Lymphoma (MK-3475-051/KEYNOTE-051)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-051; MK-3475-051 (Other: MSD Protocol Number); 2022-501257-36-00 (Registry Identifier: EU CT); U1111-1275-9516 (Registry Identifier: UTN); 2014-002950-38 (EudraCT Number)
Record Dates: First submitted 2015-01-06; First posted 2015-01-07 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Melanoma; Lymphoma; Solid Tumor; Classical Hodgkin Lymphoma; Microsatellite-instability-high Solid Tumor
Keywords: PD1; PD-1; PDL1; PD-L1; cHL; MSI-H
MeSH Terms: conditions — Melanoma; Lymphoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Melanoma (Experimental): Participants aged 6 months to <18 years with melanoma receive pembrolizumab, starting dose 2 mg/kg (maximum dose 200 mg), intravenously (IV) once every 3 weeks (Q3W). Enrollment of participants aged 6 months to <12 years with melanoma was closed with Amendment 8. Enrollment of participants aged ≥12 years to ≤18 years with melanoma continues.
  Interventions: Biological: Pembrolizumab
- Solid Tumors and Other Lymphomas (Experimental): Participants aged 6 months to <18 years with solid tumors and other lymphomas receive pembrolizumab, starting dose 2 mg/kg (maximum dose 200 mg), IV Q3W. Initial enrollment limited to programmed death-ligand 1 (PD-L1)-positive participants. PD-L1-negative participants may enroll if responses are observed. Enrollment of participants with solid tumors and other lymphomas was closed with Amendment 8.
  Interventions: Biological: Pembrolizumab
- rrcHL (Experimental): Participants aged 3 years to <18 years with rrcHL receive pembrolizumab, starting dose 2 mg/kg (maximum dose 200 mg), IV Q3W.
  Interventions: Biological: Pembrolizumab
- MSI-H (Experimental): Participants aged 6 months to <18 years with microsatellite-instability-high (MSI-H) solid tumors receive pembrolizumab, starting dose 2 mg/kg (maximum dose 200 mg), IV Q3W.
  Interventions: Biological: Pembrolizumab
- TMB-H (Experimental): Participants aged 6 months to <18 years with tumor-mutational burden-high ≥10 mutation/Mb (TMB-H) solid tumors receive pembrolizumab, starting dose 2 mg/kg (maximum dose 200 mg), IV Q3W.
  Interventions: Biological: Pembrolizumab
- Adjuvant Melanoma (Experimental): Participants aged 12 years to <18 years with resected high-risk Stage IIB, IIC, III, or IV melanoma receive pembrolizumab, starting dose 2 mg/kg (maximum dose 200 mg), intravenously (IV) once every 3 weeks (Q3W).
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475

SUMMARY:
Researchers are looking for new ways to treat children with different types of melanoma (skin cancer), solid tumors, and lymphomas (blood cancers) that are any of these:

* Advanced, which means cancer spread in the body or cannot be removed with surgery
* Relapsed, which means cancer has come back after it had responded to previous treatment (responded means it stopped growing, gets smaller, or disappeared)
* Refractory, which means cancer did not respond to previous treatment

Pembrolizumab is an immunotherapy, which is a treatment that helps the immune system fight cancer. Researchers want to learn if different doses of pembrolizumab can cause at least 1 of the types of cancer to get smaller or go away.

With Amendment 8, enrolment of participants with solid tumours and participants 6 months to under 12 years old with melanoma were closed. Enrolment of participants 12-18 years old with melanoma continues. Enrolment of participants who have tumours with specific traits (microsatellite-instability-high (MSI-H), and tumour-mutational burden-high ≥10 mutation/Mb (TMB-H)) also continues.

ELIGIBILITY:
Inclusion Criteria:

* Between 6 months and <18 years of age on day of signing informed consent is documented.
* Histologically- or cytologically-documented, locally-advanced, or metastatic solid malignancy or lymphoma that is incurable and has failed prior standard therapy, or for which no standard therapy exists, or for which no standard therapy is considered appropriate
* Any number of prior treatment regimens
* Tissue (or lymph node biopsy for rrcHL participants) available from an archival tissue sample or, if appropriate, a newly obtained core or excisional biopsy of a tumor lesion not previously irradiated
* Advanced melanoma or PD-L1-positive advanced, relapsed, or refractory solid tumor or lymphoma
* Measurable disease based on RECIST 1.1 (Or based on IWG [Cheson, 2007] [i.e., measurement must be >15 mm in longest diameter or >10 mm in short axis] for rrcHL participants)
* Participants with neuroblastoma with only metaiodobenzylguanidine (MIBG)-positive evaluable disease may be enrolled
* Lansky Play Scale ≥50 for participants from 6 months up to and including 16 years of age; or Karnofsky score ≥50 for participants >16 years of age
* Adequate organ function
* Female participants of childbearing potential should have a negative urine or serum pregnancy test within 72 hours before the first dose of study medication
* Female participant is not a woman of childbearing potential (WOCBP) or is a WOCBP who is abstinent from heterosexual intercourse or using contraception during the intervention period and for at least 120 days after the last dose of study intervention
* Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Demonstrate adequate organ function.

Exclusion Criteria:

* Currently participating and receiving study therapy in, or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the date of allocation/randomization
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the date of allocation/randomization
* Prior systemic anti-cancer therapy including investigational agent within 2 weeks prior to study Day 1 or not recovered from adverse events due to a previously administered agent
* Prior radiotherapy within 2 weeks of start of study treatment
* Known additional malignancy that is progressing or requires active treatment with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (eg, breast carcinoma, cervical carcinoma in situ) with potentially curative therapy, or in situ cervical cancer
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Tumor(s) involving the brain stem
* Severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients
* Active autoimmune disease that has required systemic treatment in past 2 years; replacement therapy (such as thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is acceptable
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Active infection requiring systemic therapy
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial through 120 days after the last dose of study medication
* Prior therapy with an anti-programmed cell death (PD)-1, anti-PD-ligand 1 (anti-PD-L1), anti-PD-L2 agent, or any agent directed to another stimulatory or inhibitory T-cell receptor (eg, cytotoxic lymphocyte associated protein-4 [CTLA-4], OX-40, CD137)
* Human immunodeficiency virus (HIV)
* Hepatitis B or C
* Known history of active tuberculosis (TB; Bacillus tuberculosis)
* Received a live vaccine within 30 days of planned start of study medication
* Has undergone solid organ transplant at any time, or prior allogeneic hematopoietic stem cell transplantation within the last 5 years. (Participants who have had an allogeneic hematopoietic transplant >5 years ago are eligible as long as there are no symptoms of Graft Versus Host Disease [GVHD].)
* History or current evidence of any condition, therapy, or laboratory abnormality, or known severe hypersensitivity to any component or analog of the trial treatment, that might confound the results of the trial, or interfere with the participant's participation for the full duration of the study
* Known psychiatric or substance abuse disorders that would interfere with the requirements of the study

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 370 (Estimated)
Dates: Start 2015-03-18 (Actual); Primary Completion 2027-10-25 (Estimated); Study Completion 2027-10-25 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors and Other Lymphoma Version 1.1 (RECIST 1.1) per Site Assessment (Each Disease Indication Evaluated Separately) | Up to 2 years
  The ORR is assessed by RECIST 1.1 per site assessment. The ORR is defined as the percentage of participants who have a response (complete response, CR or partial response, PR) prior to disease progression. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
ORR by RECIST 1.1 per Site Assessment for MSI-H or TMBH Solid Tumors (Each Cohort Evaluated Separately) | Up to 2 years
  The ORR is assessed by RECIST 1.1 per site assessment. The ORR is defined as the percentage of participants who have a response (complete response, CR or partial response, PR) prior to disease progression. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
ORR by International Working Group (IWG) Response Criteria (Cheson, 2007) per BICR Assessment for rrcHL Cohort | Up to approximately 2 years
  The ORR is assessed by blinded independent central review utilizing the International Working Group [IWG] response assessment criteria per Cheson 2007 by BICR. The ORR is defined as the percentage of participants who have a response (complete response, CR or partial response, PR) prior to disease progression. CR is the disappearance of all evidence of disease and PR is the regression of measurable disease and no new sites. Participants with missing data are considered non-responders.
Number of Participants with Dose-Limiting Toxicities (DLTs) | Cycle 1 (Up to 21 days)
  Number of participants experiencing toxicities that are possibly, probably, or definitely related to study therapy; that meet pre-defined severity criteria; and result in a change in the given dose.
Number of Participants Experiencing Adverse Events (AEs) | Up to 27 months
  An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Number of Participants Discontinuing Study Drug Due to AEs | Up to 2 years
  An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.

SECONDARY OUTCOMES:
ORR by IWG Response Criteria (Cheson, 2007) per Site Assessment (rrcHL Cohort) | Up to 2 years
  The ORR is assessed by blinded independent central review utilizing the International Working Group [IWG] response assessment criteria per Cheson 2007 by site assessment. The ORR is defined as the percentage of participants who had a response (complete response, CR or partial response, PR) prior to disease progression. CR is the disappearance of all evidence of disease and PR is the regression of measurable disease and no new sites. Participants with missing data are considered non-responders.
DOR per RECIST 1.1 by Site Assessment (Advanced Melanoma, Solid Tumors and Other Lymphoma, Each Disease Indication Is Evaluated Separately) | Up to approximately 2 years
  The duration of overall response is assessed by RECIST 1.1 by site evaluation. The duration of overall response is measured from the time measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded on study).
DOR per RECIST 1.1 by Site Assessment (MSI-H and TMBH, Each Cohort Is Evaluated Separately) | Up to approximately 2 years
  The duration of overall response is assessed by RECIST 1.1 by site evaluation. The duration of overall response is measured from the time measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded on study).
DOR per IWG 2007 (Cheson, 2007) Response by BICR Assessment (rrcHL Cohort) | Up to approximately 2 years
  The duration of overall response is measured from the time measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded on study).
DOR per IWG 2007 (Cheson, 2007) Response by Site Assessment (rrcHL Cohort) | Up to approximately 2 years
  The duration of overall response is measured from the time measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded on study).
DOR per Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST) by Site Assessment (Solid Tumors and Other Lymphoma, Each Disease Indication Evaluated Separately) | Up to approximately 2 years
  The duration of overall response is measured from the time measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded on study).
DOR per Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST) by Site Assessment (MSI-H and TMB-H, Each Cohort Is Evaluated Separately) | Up to approximately 2 years
  The duration of overall response is measured from the time measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded on study).
Progression-free Survival (PFS) Using RECIST 1.1 Criteria by Site Assessment (Solid Tumors and Other Lymphoma, Each Disease Indication Evaluated Separately) | Up to approximately 2 years
  Progression free survival is defined as the time from randomization to the first documented disease progression, or death due to any cause, whichever occurred first. PFS is assessed by using RECIST 1.1 criteria by site assessment. Median PFS will be calculated from the product-limit (Kaplan-Meier) method for censored data.
PFS using RECIST 1.1 Criteria by Site Assessment (MSI-H and TMB-H, Each Cohort Evaluated Separately) | Up to approximately 2 years
  Progression free survival is defined as the time from randomization to the first documented disease progression, or death due to any cause, whichever occurred first. PFS is assessed by using RECIST 1.1 criteria by site assessment. Median PFS will be calculated from the product-limit (Kaplan-Meier) method for censored data.
PFS using IWG 2007 Criteria (Chesson 2007) by BICR Assessment (rrcHL Cohort) | Up to approximately 2 years
  Progression free survival is defined as the time from randomization to the first documented disease progression, or death due to any cause, whichever occurred first. PFS is assessed by using IWG 2007 criteria (Chesson, 2007) by BICR assessment (rrcHL Cohort). Median PFS will be calculated from the product-limit (Kaplan-Meier) method for censored data.
PFS using IWG 2007 Criteria (Chesson, 2007) by Site Assessment (rrcHL Cohort) | Up to approximately 2 years
  Progression free survival is defined as the time from randomization to the first documented disease progression, or death due to any cause, whichever occurred first. PFS is assessed by using IWG 2007 criteria (Chesson, 2007) by site assessment. Median PFS will be calculated from the product-limit (Kaplan-Meier) method for censored data.
PFS Using irRECIST Criteria by Site Assessment | Up to approximately 2 years
  Progression free survival is defined as the time from randomization to the first documented disease progression, or death due to any cause, whichever occurred first. PFS is assessed by using irRECIST criteria by site assessment. Median PFS will be calculated from the product-limit (Kaplan-Meier) method for censored data.
Disease Control Rate by RECIST 1.1 Using Site Assessment (Solid Tumors and Other Lymphoma, Each Disease Indication Evaluated Separately) | Up to approximately 2 years
  Disease Control Rate is defined as the percentage of participants with a response of CR, PR, or SD. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study. Progressive Disease is least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Disease Control Rate by RECIST 1.1 Using Site Assessment (MSIH and TMB-H, Each Cohort Evaluated Separately) | Up to approximately 2 years
  Disease Control Rate is defined as the percentage of participants with a response of CR, PR, or SD. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study. Progressive Disease is least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Disease Control Rate by irRECIST Using Site Assessment (Solid Tumors and Other Lymphomas, Each Disease Indication Evaluated Separately) | Up to approximately 2 years
  Disease Control Rate is defined as the percentage of participants with a response of CR, PR, or SD. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study. Progressive Disease is least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Overall Survival | Up to approximately 2 years
  Overall survival is defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis will be censored at the date of the last follow-up. Median overall survival will be calculated from the product-limit (Kaplan-Meier) method for censored data.
Objective irRECIST Response Rate by Site Assessment (Each Disease Indication Evaluated Separately) | Up to approximately 2 years
  The ORR is assessed by irRECIST per site assessment.
Area Under the Concentration Curve (AUC) for Pembrolizumab | Predose Cycles 1, 2, 4, 8 and every 4 cycles thereafter, and within 30 minutes post infusion at Cycles 1 and 8. Additional single pharmacokinetic samples obtained in Cycle 1 between 72 to 168 hours post-dose, and Cycle 1 at 336 hours post-dose
  The AUC of pembrolizumab when administered as monotherapy will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (17):
- United States (7):
  - Call for Information (Investigational Site 0019), Aurora, Colorado
  - Call for Information (Investigational Site 0026), Boston, Massachusetts
  - Call for Information (Investigational Site 0031), New York, New York
  - Call for Information (Investigational Site 0070), Fargo, North Dakota
  - Call for Information (Investigational Site 0032), Cincinnati, Ohio
  - Call for Information (Investigational Site 0071), Sioux Falls, South Dakota
  - Call for Information (Investigational Site 0054), Dallas, Texas
- MSD Brasil, São Paulo, Brazil
- MSD France, Paris, France
- MSD Sharp & Dohme GmbH, München, Germany
- Merck Sharp & Dohme Co. Ltd., Hod HaSharon, Israel
- MSD Italia S.r.l., Rome, Italy
- Merck Sharp & Dohme BV, Haarlem, Netherlands
- Merck Sharp & Dohme Lda., Paço de Arcos, Portugal
- MSD Korea LTD, Seoul, South Korea
- MSD Sweden, Stockholm, Sweden
- Merck Sharp & Dohme Ltd., London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Geoerger B, Kang HJ, Yalon-Oren M, Marshall LV, Vezina C, Pappo A, Laetsch TW, Petrilli AS, Ebinger M, Toporski J, Glade-Bender J, Nicholls W, Fox E, DuBois SG, Macy ME, Cohn SL, Pathiraja K, Diede SJ, Ebbinghaus S, Pinto N. Pembrolizumab in paediatric patients with advanced melanoma or a PD-L1-positive, advanced, relapsed, or refractory solid tumour or lymphoma (KEYNOTE-051): interim analysis of an open-label, single-arm, phase 1-2 trial. Lancet Oncol. 2020 Jan;21(1):121-133. doi: 10.1016/S1470-2045(19)30671-0. Epub 2019 Dec 4. PMID 31812554
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26169&tenant=MT_MSD_9011